CLINICAL TRIAL: NCT00567541
Title: Feasibility Study of the Bioness Battery-Powered Microneuromodulator (BBPM) to Treat Chronic Shoulder Pain in Chronic Post-Stroke Subjects
Brief Title: An Implantable Microneuromodulator for the Treatment of Chronic Shoulder Pain in Chronic Post-Stroke Subjects
Acronym: BBPM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bioness Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP-BBPM-001
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Results first posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Shoulder Pain Chronic
Keywords: shoulder; pain; stroke; subluxation
MeSH Terms: conditions — Pain; Stroke; Joint Dislocations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active BBPM stimulation (Active Comparator): Therapeutic Stimulation is applied via the Battery Powered Microneuromodulator (BBPM) which is programmed to deliver set stimulation parameters with approximate frequency of 30 Hz, current 5mA for 200 microseconds for the first 12 weeks of the study. The BBPM is implanted near the axillary nerve within the quadrilateral space.
  Interventions: Device: Battery Powered Microneuromodulator (BBPM)
- Sham BBPM stimulation (Placebo Comparator): The Battery Powered Microneuromodulator is implanted near the axillary nerve within the quadrilateral space. The BBPM is programmed for the first 12 weeks of the study to deliver short bursts of extremely low amplitude electrical stimulation at very wide time intervals to give appearance, impression, and sensation of therapeutic treatment. After 24 weeks, the device will be reprogrammed to deliver therapeutic stimulation over a 12 week period.
  Interventions: Device: Battery Powered Microneuromodulator (BBPM)

INTERVENTIONS:
Device: Battery Powered Microneuromodulator (BBPM) — The Battery Powered Microneuromodulator (BBPM) is programmed to deliver bursts of electrical stimulation to deliver therapeutic stimulation beginning with a frequency of 30Hz, current of 5mA, for 200 microseconds. These settings were applied to deliver greater or lesser intensity based on study arm (active vs placebo).
  Other Names: Bioness Battery Powered Microneuromodulator

SUMMARY:
The goal of this research study is to investigate safety and gather initial effectiveness data for a new implanted device designed to treat chronic shoulder pain in chronic post-stroke subjects. The BBPM weighs less than 0.03 ounces and measures 1" x 0.1". It is implanted into the shoulder to stimulate the axillary nerve. Stimulation of this nerve may reduce shoulder pain, reduce shoulder subluxation, improve motion, improve function, and possibly decrease use of pain medication. CAUTION--Investigational device. Limited by Federal law to investigational use.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, controlled, double-blinded parallel study designed to evaluate feasibility and safety. The primary purpose of this study is to demonstrate the clinical feasibility of implanting the BBPM near a peripheral nerve for the treatment of chronic, intractable, pain in this case represented by chronic regional shoulder pain in hemiplegic stroke patients. This is a 48-week efficacy study with safety data collection throughout the study period and up to 2 years for all available subjects. Each study arm will receive therapeutic level stimulation for a total of 12 consecutive weeks (Weeks 1-12 for Active treatment group and Weeks 24-36 for the sham group) during the 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Chronic post-stroke duration greater than or equal to 6 months
* Unilateral hemiplegic shoulder pain persisting for ≥6 months
* Hemiparesis (shoulder abduction graded <5/5 on Manual Muscle Testing ipsilateral to the shoulder in which the subject has chronic pain
* Shoulder pain ≥ 6/10 (on 0-10 numeric rating scale (NRS) for worst pain in last week (BPI #12))
* Ability to give informed consent and understand study requirements
* Ability to quantify pain using a 0-10 numeric rating scale. (A screening tool will be used to ensure that participants can rate 3 common pain scenarios (mosquito bite, stubbed toe and broken bone) on a 0-10 NRS relative to each other.)
* Willing and able to understand and comply with all study-related procedures during the course of the study
* Motivated to maintain an accurate diary for the study duration

Exclusion Criteria:

* Hemineglect (i.e., extinguish to double simultaneous stimulation)
* Shoulder trauma or diagnosed shoulder pathology prior to stroke; history of any shoulder surgery, regardless of whether procedure preceded for followed stroke.
* Need to take >1 pain medication (opioid or non-opioid) for shoulder pain
* Regular use of pain medication for chronic pain other than shoulder pain
* Anticoagulated (taking warfarin or heparin, including fractionated heparin) or has a bleeding disorder
* Unable, per their prescribing physician, to stop antiplatelet medications (e.g., aspirin, ticlopidine (Ticlid), clopidogrel (Plavix), tirofiban (Aggrastat), and eptifibatide (Integrilin)) for at least 7 days prior to device implantation.
* Cardiac pacemaker
* Implanted neurostimulator (e.g., spinal cord, deep brain, vagus nerve) or implanted pump or infusion device
* Prosthetic heart valve or valvular heart disease requiring antibiotic prophylaxis
* History of cardiac arrhythmia with hemodynamic instability
* Uncontrolled seizures (> 1 seizure per month)
* Pregnant or plan on becoming pregnant during the study period
* Medical instability
* Currently require, or likely to require, diathermy
* Currently require, or anticipated to require, MRI within 8 weeks of projected device implantation date
* History of adverse reactions to local anesthetic (e.g., lidocaine)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-06; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Friedman, MD, Principal Investigator — Virginia Mason Seattle Main Clinic; Tim Deer, MD, Principal Investigator — The Center for Pain Relief; Ziyad Ayyoub, M.D., Principal Investigator — Rancho Los Amigos National Rehabilitation Center
Locations (3):
- United States (3):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - Virginia Mason Medical Center, Seattle, Washington
  - The Center for Pain Relief, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active BBPM Stimulation: The Battery Powered Microneuromodulator (BBPM) is programmed to deliver set therapeutic stimulation parameters for the first 12 weeks of the study.
  Battery Powered Microneuromodulator (BBPM): The Battery Powered Microneuromodulator (BBPM) will be programmed for the first 12 weeks of the study to deliver therapeutic amplitude electrical stimulation. therapeutic treatment.
- Sham BBPM Stimulation: The Battery Powered Microneuromodulator(BBPM) will be programmed for the first 12 weeks of the study to deliver short bursts of extremely low amplitude electrical stimulation at very wide time intervals to give appearance, impression, and sensation of therapeutic treatment. After 24 weeks, they will be reprogrammed to receive therapeutic stimulation.
  Battery Powered Microneuromodulator (BBPM): The Battery Powered Microneuromodulator (BBPM) is programmed for the first 12 weeks of the study to deliver short bursts of extremely low amplitude electrical stimulation at very wide time intervals to give appearance, impression, and sensation of therapeutic treatment. After 24 weeks, the device will be reprogrammed to deliver therapeutic stimulation.
Period: Overall Study
Arm/Group | Active BBPM Stimulation | Sham BBPM Stimulation
Started | 7 | 9
Completed | 7 | 8
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: fifteen of 16 subjects were randomized and their devices activated. One subject experienced and AE prior to device activation and was exited from the study
Groups:
- Active BBPM Stimulation: Active Battery Powered Microneuromodulator (BBPM): The Battery Powered Microneuromodulator (BBPM) is programmed for the first 12 weeks of the study to deliver therapeutic amplitude electrical stimulation.
- Sham BBPM Stimulation: Sham Battery Powered Microneuromodulator (BBPM): The Battery Powered Microneuromodulator (BBPM) is programmed for the first 12 weeks of the study to deliver short bursts of extremely low amplitude electrical stimulation at very wide time intervals to give appearance, impression, and sensation of therapeutic treatment. After 24 weeks, the device will be reprogrammed to deliver therapeutic stimulation.
- Total: Total of all reporting groups
Arm/Group | Active BBPM Stimulation | Sham BBPM Stimulation | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Customized [Number; unit: participants]
  35-55 years old | 1 | 3 | 4
  56-80 years old | 6 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 5 | 3 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  white | 5 | 7 | 12
  non-white | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Relief of Chronic Shoulder Pain
Description: Brief Pain Inventory (BPI) Question # 12 (rating pain at its worst in week prior to visit) was used to measure number of participants in whom BBPM provided any relief from chronic shoulder pain after implantation, as evidence by appropriate muscular contraction and/or paresthesia. BPI scale range is from 1 to 10, where 0 = 'no pain' and 10 = 'pain as bad as one can imagine'.
Time Frame: From baseline to 48 week follow up
Population: Intent to Treat population was analyzed
Measure: Number; unit: participants
Groups:
- Active BBPM Stimulation: The.Battery Powered Microneuromodulator (BBPM): The Battery Powered Microneuromodulator (BBPM) is programmed for the first 12 weeks of the study to deliver therapeutic amplitude electrical stimulation.
- Sham BBPM Stimulation: The Battery Powered Microneuromodulator (BBPM): The Battery Powered Microneuromodulator (BBPM) is programmed for the first 12 weeks of the study to deliver short bursts of extremely low amplitude electrical stimulation at very wide time intervals to give appearance, impression, and sensation of therapeutic treatment. After 24 weeks, the device is reprogrammed to deliver therapeutic stimulation.
Arm/Group | Active BBPM Stimulation | Sham BBPM Stimulation
Number analyzed (Participants) | 7 | 9
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout trial up to one year
Arm/Group | Active BBPM Stimulation | Sham BBPM Stimulation
Serious Adverse Events (participants affected / at risk) | 2/7 | 6/9
Other Adverse Events (participants affected / at risk) | 7/7 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active BBPM Stimulation (N=7) | Sham BBPM Stimulation (N=9)
Ischemic Stroke (Nervous system disorders) | 1 (1) | 4 (4) — non-device related
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — non-device related
bone fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — non-device related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active BBPM Stimulation (N=7) | Sham BBPM Stimulation (N=9)
Implant site pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — device related
Increased pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — device related
Pain other than at implant site (General disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) — device related
Device Migration (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) — device related
Collateral Muscle Stimulation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — device related
Edema/Swelling (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) — device related
Migraine (Nervous system disorders) | 1 (1) | 3 (3) — non-device related
fall (Nervous system disorders) | 4 (4) | 1 (1) — non-device related
Nausea, vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) — non-device related
Flu, shingles (Infections and infestations) | 1 (1) | 1 (1) — non-device related
general complaints (General disorders) | 3 (3) | 6 (6) — non-device related
Spasticity, hang grip issues (Nervous system disorders) | 2 (2) | 3 (3) — non-device related

LIMITATIONS AND CAVEATS:
Further study plans terminated due to high migration/adverse event rates Small sample size Didn't include socio-environmental factors which could affect subject's overall functionality Three different sites/subtle stimulator implantation variances

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less